CLINICAL TRIAL: NCT02755441
Title: Pulmonary Fibrosis Biomarker Cohort (PFBIO)
Brief Title: Pulmonary Fibrosis Biomarker Cohort - a Prospective Cohort of Incident Patients With IPF
Acronym: PFBIO
Status: Active, not recruiting | Type: Observational
Sponsor: Nils Hoyer (Other)
Collaborators: Aarhus University Hospital (Other); Nordic Bioscience A/S (Industry)
Responsible Party: Sponsor-Investigator, Nils Hoyer, MD, University Hospital, Gentofte, Copenhagen
Organization: University Hospital, Gentofte, Copenhagen (Other)
Other Study IDs: PFBIO
Record Dates: First submitted 2016-04-19; First posted 2016-04-29 (Estimated); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Diagnosis; Prognosis; Biomarker
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and EDTA-plasma is collected from all patients at 0, 6 and 12 months, 2 years, 3 years, 4 years and 5 years.
  Blood DNA and RNA tubes are collected for all patients at one site (Gentofte hospital)
Oversight: Data Monitoring Committee: No

SUMMARY:
Incident patients with idiopathic pulmonary fibrosis (IPF) in Denmark will be offered inclusion and followed up for up to 5 years with measurements of blood biomarkers and measurements of disease progression.

DETAILED DESCRIPTION:
IPF pathogenesis is complex, including epithelial injury, resident fibroblast-myofibroblast transformation, recruitment of fibrocytes, macrophage activation, and release of numerous cytokines and chemokines. Several of these processes release potential biomarker proteins into the blood stream or onto the epithelial surface where they can be measured. Biomarkers have mainly two potential roles in IPF. Firstly, a diagnostic biomarker would distinguish IPF from other diseases with similar symptoms, facilitating diagnosis and possibly decreasing the need for risky procedures, such as surgical lung biopsy. Secondly, a prognostic biomarker would distinguish rapid progressors from slow progressors, which is difficult today.

This study will prospectively include patients at the two largest centres in Denmark where patients are treated for IPF and has thus a good opportunity to include the majority of incident cases of IPF in Denmark. The blood levels of several promising biomarkers will be measured at baseline and during up to 5 years follow-up. Patients will also be followed up through regular clinical examination and by querying national registries to determine disease progression, mortality, healthcare utilization and selected co-morbidities. The database will be used for determination of risk factors for the outcomes listed above. Sub-group analyses are planned in respect to sex, treatment, radiologic imaging, smoking status, clinical data such as pulmonary function tests, co-morbidities (both pulmonary disease and extra-pulmonary disease), and disease severity at baseline.

A research biobank with blood samples is established from the study population. This biobank, and the database of newly diagnosed IPF patients, will be used for future research in IPF.

The prospectively created database will also be used for future research in IPF.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic pulmonary fibrosis according to the 2011 guidelines by the American Thoracic Cosicety (ATS) and European Respiratory Society (ERS)

Exclusion Criteria:

* Age lower than 18 years
* Unable to provide informed consent to participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Incidental patients diagnosed with idiopathic pulmonary fibrosis (IPF) at Gentofte hospital and Aarhus university hospital are screened for inclusion
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2016-04; Primary Completion 2023-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Disease progression or mortality | 1 year
  Number of patients who fulfil any of the following: disease progression or death

SECONDARY OUTCOMES:
Hospitalizations | 1 year
  Number of respiratory and non-respiratory hospitalizations
Exacerbations | 1 year
  Number of acute exacerbations of idiopathic pulmonary fibrosis
Lung function tests | 1 year
  Reduction in diffusion capacity (DLCO) and forced vital capacity (FVC)
Mortality | 1 year
  All-cause and disease-specific mortality
Change in quality of life | 1 year
  Change in St. George Respiratory Questionnaire, symptom scores
Combined end-point of disease progression | 1 year
  Number of patients who fulfill any of the following: decrease in lung function, reduced walking distance at 6 minutes walking test, increased need for supplementary oxygen, hospitalization
Progression in serum/plasma biomarker levels | 1 year
  Increase or decrease in serum/plasma biomarker levels.

CONTACTS AND LOCATIONS:
Overall Officials: Nils Hoyer, MD, Principal Investigator — Gentofte Hospital
Locations (2):
- Denmark (2):
  - Gentofte Hospital, Hellerup, Copenhagen
  - Aarhus University Hospital, Aarhus

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Raghu G, Collard HR, Egan JJ, Martinez FJ, Behr J, Brown KK, Colby TV, Cordier JF, Flaherty KR, Lasky JA, Lynch DA, Ryu JH, Swigris JJ, Wells AU, Ancochea J, Bouros D, Carvalho C, Costabel U, Ebina M, Hansell DM, Johkoh T, Kim DS, King TE Jr, Kondoh Y, Myers J, Muller NL, Nicholson AG, Richeldi L, Selman M, Dudden RF, Griss BS, Protzko SL, Schunemann HJ; ATS/ERS/JRS/ALAT Committee on Idiopathic Pulmonary Fibrosis. An official ATS/ERS/JRS/ALAT statement: idiopathic pulmonary fibrosis: evidence-based guidelines for diagnosis and management. Am J Respir Crit Care Med. 2011 Mar 15;183(6):788-824. doi: 10.1164/rccm.2009-040GL. PMID 21471066
- [Derived] Hoyer N, Prior TS, Bendstrup E, Shaker SB. Diagnostic delay in IPF impacts progression-free survival, quality of life and hospitalisation rates. BMJ Open Respir Res. 2022 Jul;9(1):e001276. doi: 10.1136/bmjresp-2022-001276. PMID 35798532